CLINICAL TRIAL: NCT05631327
Title: Phase 1, Open-Label, Dose-Finding, and Expansion Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Activity of JZP341 in Adult Participants With Advanced or Metastatic Solid Tumors
Brief Title: A JZP341 Study in Adult Participants With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated based on a business decision by the Sponsor.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JZP341-102
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: Advanced Solid Tumor; Metastatic Solid Tumor; JZP341
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Finding Phase: JZP341 (Experimental): Participants who will receive JZP341 on Day 1 and Day 15 of each 28-day cycle.
  Interventions: Drug: JZP341
- Dose Expansion Phase: JZP341 (Experimental): Participants who will receive JZP341 at the RP2D established in the Dose Finding Phase on Day 1 and Day 15 of each 28-day cycle.
  Interventions: Drug: JZP341

INTERVENTIONS:
Drug: JZP341 — JZP341 will be administered as a single, intravenous infusion over 2 hours.

SUMMARY:
This study will assess the safety and efficacy of JZP341 in participants with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, multiple-dose, phase 1, multicenter, dose-finding study of single-agent JZP341 followed by a targeted expansion phase.

This study will have 2 phases: Dose Finding Phase and Dose Expansion Phase.

The Dose-Finding Phase will determine the recommended phase 2 dose (RP2D), assess safety and pharmacokinetics/pharmacodynamics, and explore preliminary antitumor activity of JZP341 in participants with relapsed or refractory advanced solid tumors.

The Dose-Expansion Phase will evaluate clinical activity and further evaluate the safety of multiple doses of single-agent JZP341 at the RP2D in participants with relapsed or refractory colorectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF)
* ≥ 18 years of age at the time of signing the ICF
* Eastern Cooperative Oncology Group performance status of 0 to 2
* Adequate bone marrow reserve
* Adequate coagulation function, liver/pancreas function, and renal function
* No clinically significant abnormalities in the levels of serum electrolytes
* Life expectancy >12 weeks
* Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 3 months after the last dose of study intervention:

  * Refrain from donating sperm, AND either:
  * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent, OR
  * Must agree to use an approved contraception method
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Woman of non-childbearing potential (WONCBP)
  * Woman of childbearing potential (WOCBP) and using an effective contraceptive method
* A WOCBP must have a negative highly sensitive pregnancy test within 72 hours of the first dose of study intervention

Inclusion Criteria for Dose Finding Phase Only:

* Have a histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumor that has progressed after prior standard therapy, been intolerant to or is ineligible for standard therapy, or has a malignancy for which there is no approved therapy considered standard of care

Inclusion Criteria for Dose Expansion Phase Only:

* Histologically or cytologically confirmed colorectal adenocarcinoma that has progressed on or is intolerant to treatment from fluoropyrimidine, oxaliplatin, and irinotecan. Participants may have received bevacizumab, anti-epidermal growth factor receptor monoclonal antibody, or checkpoint inhibitor as appropriate.
* Measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 criteria

Exclusion Criteria:

* Primary central nervous system (CNS) tumor or symptomatic CNS metastases that are neurologically unstable or have required increasing doses of steroids within the 4 weeks prior to study entry to manage CNS symptoms (symptomatic brain metastases that have been adequately treated are not excluded)
* Any clinically significant cardiac disease defined as New York Heart Association class III or IV within the 6 months before Screening
* History of ≥ Grade 3 pancreatitis
* History of intracranial thrombosis or history of recurrent thrombosis (except for catheter-related thrombosis)
* Active (significant or uncontrolled) gastrointestinal bleeding
* Active uncontrolled infection (≥ Grade 2) at the time of enrollment
* HIV-positive, unless:

  * CD4+ count ≥ 300/μL;
  * Undetectable viral load; AND
  * Receiving highly active antiretroviral therapy
* Uncontrolled infection of hepatitis B or hepatitis C or diagnosis of immunodeficiency

  * Participants with Hepatitis B who have controlled infection are permitted. Participants with controlled infections must undergo periodic monitoring of Hepatitis B virus DNA. Participants must remain on antiviral therapy for ≥ 6 months beyond the last dose of study intervention.
* Pregnant (or plan to be pregnant) or lactating woman
* History of any severe or uncontrolled medical condition
* Unresolved toxicity, based on the investigator's assessment of the participant, from prior radiation, chemotherapy, or other targeted treatment, including investigational treatment, except for stable conditions ≤Grade 2 (ie, neuropathy, myalgia, fatigue, alopecia, therapy-related endocrinopathies)
* Prior treatment with JZP341 or any other asparaginase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose-Limiting Toxicities (Dose Finding Phase) | Baseline up to Day 28
Number of Participants With Treatment-emergent Adverse Events, by Severity (Dose Finding and Dose Expansion Phases) | Baseline up to 5 years
Pharmacokinetic Parameter Area Under the Concentration-Time Curve (AUC) of JZP341 (Dose Finding Phase) | Cycle 1 Day (Dy) 1: (pre & post-dose, 4 hour [hr], 8hr), Dys 2,3,4,8,11,15 (pre & post-dose),22,29; Cycle 2 Dy 1 (pre & post-dose, 8hr), Dys 4,8,15 (pre & post-dose), 29; Cycle 3+, Dys 1 (pre & post-dose), 4hr (Cycle 3 only), and 15 (each cycle, 28 dys)
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) Levels of JZP341 (Dose Finding Phase) | Cycle 1 Day (Dy) 1: (pre & post-dose, 4 hour [hr], 8hr), Dys 2,3,4,8,11,15 (pre & post-dose),22,29; Cycle 2 Dy 1 (pre & post-dose, 8hr), Dys 4,8,15 (pre & post-dose), 29; Cycle 3+, Dys 1 (pre & post-dose), 4hr (Cycle 3 only), and 15 (each cycle, 28 dys)
Pharmacokinetic Parameter Time to Maximum Plasma Concentration (Tmax) of JZP341 (Dose Finding Phase) | Cycle 1 Day (Dy) 1: (pre & post-dose, 4 hour [hr], 8hr), Dys 2,3,4,8,11,15 (pre & post-dose),22,29; Cycle 2 Dy 1 (pre & post-dose, 8hr), Dys 4,8,15 (pre & post-dose), 29; Cycle 3+, Dys 1 (pre & post-dose), 4hr (Cycle 3 only), and 15 (each cycle, 28 dys)
Pharmacokinetic Parameter Apparent Terminal Elimination Half-life (t1/2) of JZP341 (Dose Finding Phase) | Cycle 1 Day (Dy) 1: (pre & post-dose, 4 hour [hr], 8hr), Dys 2,3,4,8,11,15 (pre & post-dose),22,29; Cycle 2 Dy 1 (pre & post-dose, 8hr), Dys 4,8,15 (pre & post-dose), 29; Cycle 3+, Dys 1 (pre & post-dose), 4hr (Cycle 3 only), and 15 (each cycle, 28 dys)
Pharmacokinetic Parameter Clearance (CL) of JZP341 (Dose Finding Phase) | Cycle 1 Day (Dy) 1: (pre & post-dose, 4 hour [hr], 8hr), Dys 2,3,4,8,11,15 (pre & post-dose),22,29; Cycle 2 Dy 1 (pre & post-dose, 8hr), Dys 4,8,15 (pre & post-dose), 29; Cycle 3+, Dys 1 (pre & post-dose), 4hr (Cycle 3 only), and 15 (each cycle, 28 dys)
Pharmacokinetic Parameter Volume of Distribution (Vd) of JZP341 (Dose Finding Phase) | Cycle 1 Day (Dy) 1: (pre & post-dose, 4 hour [hr], 8hr), Dys 2,3,4,8,11,15 (pre & post-dose),22,29; Cycle 2 Dy 1 (pre & post-dose, 8hr), Dys 4,8,15 (pre & post-dose), 29; Cycle 3+, Dys 1 (pre & post-dose), 4hr (Cycle 3 only), and 15 (each cycle, 28 dys)
Nadir Serum Asparaginase Activity Response Rate (Dose Finding Phase) | Baseline up to Day 14
  Nadir serum asparaginase activity (NSAA) response rate is defined as the proportion of participants achieving NSAA ≥ 0.1 U/mL at 14 days following the first dose of JZP341 administration.
Disease Control Rate (Dose Expansion Phase) | Baseline up to Week 12

SECONDARY OUTCOMES:
Proportion of Participants With Hypersensitivity Reactions, Anti-Drug Antibodies, and Neutralizing Antibodies (Dose Finding and Dose Expansion Phases) | Baseline up to 60 days after last dose
Pharmacodynamic Parameter Change From Baseline in Plasma Glutamine Concentrations (Dose Finding and Dose Expansion Phases) | Cycle 1 Day (Dy) 1: (pre&post, 4 hour [hr], 8hr), Dys 2&3 (DFP), 4,8,11 (DFP), 15 (pre&post), 22 (DFP), 29; Cycle 2, Dy 1:pre&post, 8hr (DFP), Dys 4&8 (DFP), 15 pre, 15 post (DFP); Cycle 3+:Dy1 pre&post, 4 hr (Cycle 3 DFP only), 15 (each cycle, 28 days)
Pharmacodynamic Parameter Change From Baseline in Plasma Asparagine Concentrations (Dose Finding and Dose Expansion Phases) | Cycle 1 Day (Dy) 1: (pre&post, 4 hour [hr], 8hr), Dys 2&3 (DFP), 4,8,11 (DFP), 15 (pre&post), 22 (DFP), 29; Cycle 2, Dy 1:pre&post, 8hr (DFP), Dys 4&8 (DFP), 15 pre, 15 post (DFP); Cycle 3+:Dy1 pre&post, 4 hr (Cycle 3 DFP only), 15 (each cycle, 28 days)
Serum Asparaginase Activity of JZP341 (Dose Expansion Phase) | Cycle 1, Dose 1: predose; Cycle 1, Dose 2: predose; Cycle 2 and subsequent cycles: predose on Day 1 of each cycle and at the 60-day follow-up visit (each cycle is 28 days)
Pharmacokinetic Parameter Area Under the Concentration-Time Curve (AUC) of JZP341 (Dose Expansion Phase) | Cycle 1 Day 1 [pre- and post-dose, 4hour (hr), 8hr], Days 4, 8, 15 (pre- and post-dose) and 29; Cycle 2+: Days 1 (pre and post) and 15, and if last dose, Days 22 and 29 (each cycle, 28 days)
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) Levels of JZP341 (Dose Expansion Phase) | Cycle 1 Day 1 [pre- and post-dose, 4hour (hr), 8hr], Days 4, 8, 15 (pre- and post-dose) and 29; Cycle 2+: Days 1 (pre and post) and 15, and if last dose, Days 22 and 29 (each cycle, 28 days)
Pharmacokinetic Parameter Time to Maximum Plasma Concentration (Tmax) of JZP341 (Dose Expansion Phase) | Cycle 1 Day 1 [pre- and post-dose, 4hour (hr), 8hr], Days 4, 8, 15 (pre- and post-dose) and 29; Cycle 2+: Days 1 (pre and post) and 15, and if last dose, Days 22 and 29 (each cycle, 28 days)
Pharmacokinetic Parameter Apparent Terminal Elimination Half-life (t1/2) of JZP341 (Dose Expansion Phase) | Cycle 1 Day 1 [pre- and post-dose, 4hour (hr), 8hr], Days 4, 8, 15 (pre- and post-dose) and 29; Cycle 2+: Days 1 (pre and post) and 15, and if last dose, Days 22 and 29 (each cycle, 28 days)
Pharmacokinetic Parameter Clearance (CL) of JZP341 (Dose Expansion Phase) | Cycle 1 Day 1 [pre- and post-dose, 4hour (hr), 8hr], Days 4, 8, 15 (pre- and post-dose) and 29; Cycle 2+: Days 1 (pre and post) and 15, and if last dose, Days 22 and 29 (each cycle, 28 days)
Pharmacokinetic Parameter Volume of Distribution (Vd) of JZP341 (Dose Expansion Phase) | Cycle 1 Day 1 [pre- and post-dose, 4hour (hr), 8hr], Days 4, 8, 15 (pre- and post-dose) and 29; Cycle 2+: Days 1 (pre and post) and 15, and if last dose, Days 22 and 29 (each cycle, 28 days)
Nadir Serum Asparaginase Activity Response Rate (Dose Expansion Phase) | Baseline up to Day 14
  Nadir serum asparaginase activity (NSAA) response rate is defined as the proportion of participants achieving NSAA ≥ 0.1 U/mL at 14 days following the first dose of JZP341 administration.
Disease Control Rate (Dose Finding Phase) | Baseline up to Week 12
Objective Response Rate as Assessed By the Investigator (Dose Finding and Dose Expansion Phases) | Baseline and then every 6 weeks from Cycle 1 Day 1 until disease progression for 24 weeks, then every 8 weeks thereafter until disease progression, withdrawal of consent, new therapy, or death (each cycle 28 days), whichever occurs first, up to 1 year
Duration of Response as Assessed By the Investigator (Dose Finding and Dose Expansion Phases) | Baseline and then every 6 weeks from Cycle 1 Day 1 until disease progression for 24 weeks, then every 8 weeks thereafter until disease progression, withdrawal of consent, new therapy, or death (each cycle 28 days), whichever occurs first, up to 1 year
Progression-free Survival (Dose Expansion Phase) | Baseline and then every 6 weeks from Cycle 1 Day 1 until disease progression for 24 weeks, then every 8 weeks thereafter until disease progression, withdrawal of consent, new therapy, or death (each cycle 28 days), whichever occurs first, up to 1 year
Overall Survival (Dose Expansion Phase) | Baseline and then every 6 weeks from Cycle 1 Day 1 until disease progression for 24 weeks, then every 8 weeks thereafter until disease progression, withdrawal of consent, new therapy, or death (each cycle 28 days), whichever occurs first, up to 1 year

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - SCRI HealthOne, Denver, Colorado
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Oklahoma University- Oklahoma City, Oklahoma City, Oklahoma
  - Thomas Jefferson University/Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology - Nashville, Nashville, Tennessee